CLINICAL TRIAL: NCT03106441
Title: PREOPTI-POOP: Preoxygenation Optimisation in Obese Patients: High-flow Nasal Cannula Oxygen Versus Non-invasive Ventilation : A Single-centre Randomized Controlled Study. "
Brief Title: Preoxygenation Optimisation in Obese Patients
Acronym: PREOPTI-POOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC17_0046
Record Dates: First submitted 2017-03-28; First posted 2017-04-10 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Severe Obesity Design as BMI > 35kg/m2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High flow oxygen therapy by nasal cannula (Experimental): Experimental Device : High flow oxygen therapy by nasal cannula.
  Interventions: Device: High flow oxygen therapy by nasal cannula. Optiflow®
- Facial mask oxygenation in BIPAP ventilation (Active Comparator): Active Comparator: Facial mask oxygenation in BIPAP ventilation
  Interventions: Device: Facial mask oxygenation in BIPAP ventilation

INTERVENTIONS:
Device: High flow oxygen therapy by nasal cannula. Optiflow® — Patients randomized in interventional group will received a four minutes preoxygenation period with High Flow nasal cannula (60 l/mn FiO2 = 1) before orotracheal intubation. The device will be maintained in place throughout the intubation procedure in order to achieve apnoeic oxygenation.
  Arms: High flow oxygen therapy by nasal cannula
Device: Facial mask oxygenation in BIPAP ventilation — Patients randomized in BIPAP group will receive a four minutes preoxygenation with EPAP 5, IPAP 15 FiO2 = 1 for a pressure support of 10 cm H2O. The facial mask with be removed after before crash induction enabling laryngoscopic vision
  Arms: Facial mask oxygenation in BIPAP ventilation

SUMMARY:
Oro-tracheal intubation in operating room in obese patients with BMI > 35kg/m2 remains a critical event. The aim of this study is to determine whether Nasal High Flow Therapy by nasal cannula Optiflow® is more efficient than the BIPAP preoxygenation before orotracheal intubation after crash induction in obese patients

DETAILED DESCRIPTION:
This study will be designed as followed : Patients will be randomized in 2 groups :

* Preoxygenation during 4 minutes with High Flow Nasal Cannula (60l/min FiO2 (fraction of inspired oxygen) = 1) before orotracheal intubation after crash induction. The device will be maintained in place throughout the intubation procedure in order to achieve apnoeic oxygenation.
* Or Preoxygenation during 4 minutes with Bi-level Positive Airway Pressure (BIPAP) with Expiratory Positive Airway Pressure (EPAP) + 5 cm H2O and Inspiratory Airway Positive Airway Pressure (IPAP) + 15, meaning a 10cm H2O pressure support. The facial mask with be removed after before crash induction enabling laryngoscopic vision.

ELIGIBILITY:
Inclusion Criteria:

* Obese patient with BMI > 35kg/m2
* Age between 18 and 80 years
* Requiring a crash induction sequence for oro-tracheal intubation.

Exclusion Criteria:

* Pulse oxymetry < 90% in ambient air
* Haemodynamic instability
* Burned patient
* Indication of intubation vigil in spontaneous ventilation
* Patients with a documented Cormack IV exposition before inclusion
* Protected adult
* Pregnancy
* Lack of consent
* Patient already enrolled in an other randomized study looking forward improving preoxygenation quality.
* Lack of French social protection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Expired fraction of oxygen at the end of intubation | 2 minutes
  To determine whether High-Flow nasal cannula used during the preoxygenation in obese patient is more efficient than BIPAP preoxygenation.

SECONDARY OUTCOMES:
Improvement of quality of preoxygenation | 4 minutes
  duration of proceedings
Reduction in side effects incidence related to intubation | 1 hour
  Notification of adverse events during the intubation period
morbi-mortality during surgery | 6 hour
  Per and postoperative complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Karim Asehnoune, PHD, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Hôtel Dieu, Medical intensive care unit, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vourc'h M, Baud G, Feuillet F, Blanchard C, Mirallie E, Guitton C, Jaber S, Asehnoune K. High-flow Nasal Cannulae Versus Non-invasive Ventilation for Preoxygenation of Obese Patients: The PREOPTIPOP Randomized Trial. EClinicalMedicine. 2019 Jun 5;13:112-119. doi: 10.1016/j.eclinm.2019.05.014. eCollection 2019 Aug. PMID 31528849